CLINICAL TRIAL: NCT04649047
Title: Weight Loss Intervention for Mothers With Young Children
Brief Title: Lifestyle Behavior Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Mei-Wei Chang, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020B0322
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Weight Loss
Keywords: low-income women; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be assigned to the experimental group and receive a 3-weekly intervention via web and individual health coaching. The educational topics cover stress management, healthy eating, and physical activity
  Interventions: Behavioral: Goal-oriented episodic future thinking

INTERVENTIONS:
Behavioral: Goal-oriented episodic future thinking — All participants will receive a 3-week web-based intervention plus individual health coaching. The intervention topics include stress management, healthy eating, and physical activity

SUMMARY:
This lifestyle behavior intervention aims to weight loss in low-income overweight or obese mothers of young children through promotion of stress management, healthy eating, and physical activity. All eligible women will be assigned to the intervention group. The intervention will last 3 weeks and will be delivered via weekly web and individual health coaching sessions.

DETAILED DESCRIPTION:
Previous research in lifestyle behavior weight loss intervention has 3 limitations. (1) Low-income overweight or obese mothers of young children have been significantly underrepresented. (2) Prior lifestyle interventions in overweight or obese mothers have suffered from threats to internal validity and have not specifically addressed motivation, emotion, and cognition (especially executive function), all of which are critical for promoting and maintaining healthy lifestyle behaviors and health outcomes. (3) There has been little evidence that any of the potentially efficacious strategies researched previously were even possible under real-world conditions. The proposed small pilot study builds on strength and effectively addresses limitations of prior research. The ultimate goal of the proposed study is to create a more feasible and scalable intervention that can be easily implemented and sustained in real-world settings. This self-directed, web-based goal-oriented episodic future thinking intervention will focus on increasing motivation (autonomous motivation and self-efficacy) and improving emotion (emotion control and stress) and cognition (impulsivity). the will lead to weight loss and decrease risk of chronic conditions associated with obesity, for example, hypertension, type 2 diabetes, and cancer. All eligible women will be assigned to the intervention group. The intervention will last 3 weeks and will be delivered via weekly web and individual health coaching sessions. We will enroll 30 low-income overweight or obese mothers of young children with diverse racial and ethnic backgrounds. All participants will be assessed at baseline (T1) and immediately after the three-week intervention (T2). Specific aims are to to (1) assess intervention fidelity (dose, delivery, receipt) and acceptability by the study participants, (2) investigate potential intervention impact on the primary (body weight) and secondary outcomes (waist circumference), (3) explore potential intervention impact on lifestyle behaviors (diet and physical activity), (4) explore potential intervention impact on motivation (autonomous motivation, self-efficacy, social support), emotion (emotion control, stress), and cognition (impulsivity), and (5) assess cost of different recruitment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25.0-39.9 kg/m2 (calculated using height and weight)
* Current enrollment in government assistant programs (for example, WIC, food stamp (SNAP), or Madicaid)
* 6 weeks - 3.5 years postpartum
* 18-45 years old
* Fluency in speaking, reading, and writing English
* Ownership of a smart phone with unlimited text messages and internet access
* Committed to a three-week intervention study

Exclusion Criteria:

* Current pregnancy or lactation
* Plan to become pregnant during the trial
* Type 1 or 2 diabetes
* Untreated thyroid disease
* Drug or alcohol abuse or dependence within last six months
* Major psychiatric disorder (e.g., schizophrenia, bipolar)
* History of bulimia or anorexia
* Current taking of appetite suppressant or (antipsychotic) medications known to affect body weight
* Current participation in a weight control or drug study
* Current or planned participation in a commercial weight loss program
* Previous weight loss surgery
* Contraindications to physical activity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be a mother young children
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Wei Chang, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 15
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Marital Status [Count of Participants; unit: Participants]
  Single (never married) | 8
  Married | 5
  Divorced | 2
Education [Count of Participants; unit: Participants]
  High School/GED | 1
  Some College/Technical School (no degree) | 5
  Associate's Degree | 1
  Bachelor's Degree | 4
  Master's Degrees. | 4
Employment [Count of Participants; unit: Participants]
  Full-Time | 4
  Part-Time | 3
  Self-Employed | 1
  Not employed outside of home | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Self-reported body weight
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Intervention
Number analyzed (Participants) | 12
pounds
  T1 (baseline) | 194.1 (38.04)
  T2 (post-intervention) | 191.2 (37.70)
  T2 vs. T2 | -2.92 (4.23)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.036, t-test, 2 sided; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-5.6 to -0.23]

2. Secondary Outcome: Body Mass Index
Description: kg/m^2
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Intervention
Number analyzed (Participants) | 12
kg/m2
  T1 (baseline) | 32.14 (5.23)
  T2 (post-intervention) | 31.58 (5.20)
  Change from T1 to T2 | -.56 (.73)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = -0.77, t-test, 2 sided; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.02 to -0.10]

3. Secondary Outcome: Daily Dietary Fat Intake
Description: NCI brief dietary fat intake survey was used to measure dietary fat intake. Participants reported the frequency of each specific food eaten over the past 12 months. Values are:1 = never, 2 = less than once per month,3 = 1-3 times per week, 4 = 3-4 times per week,5 = 5-6 times per week, 6 = 1 time per day, 7 = 2 or more times per day. Higher scores indicate more frequent fat intake.There is no minimum or maximum available for this measure.
  The following procedures were used to convert an individual's responses to an estimate of that individual's percentage energy from fat: The frequency reported categorically on the questionnaire was converted to the number of times fat was consumed per day as shown below. In general, the midpoint of the frequency range was used.
  Never 0.0 Less than once a month 0.018 1-3 times per month 0.066 1-2 times per week 0.214 3-4 times per week 0.499 5-6 times per week 0.784
  1. time per day 1.0
  2. or more times per day 2.0
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: Times fat consumed per day
Arm/Group | Intervention
Number analyzed (Participants) | 12
Times fat consumed per day
  T1 (baseline) | 34.59 (4.93)
  T2 (post-intervention) | 31.17 (5.06)
  T2 vs. T1 | -3.42 (6.72)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = -0.51, t-test, 2 sided; Mean Difference (Final Values) = -3.42, 95% CI 2-sided [-7.69 to 0.85]

4. Secondary Outcome: Daily Fruit and Vegetable Intake
Description: NCI brief Fruit and Vegetable intake survey was used to measure dietary intake. Participants reported the frequency of each specific food eaten over the past 12 months. Values are:1 = never, 2 = less than once per month,3 = 1-3 times per week, 4 = 3-4 times per week,5 = 5-6 times per week, 6 = 1 time per day, 7 = 2 or more times per day. Higher scores indicate more frequent fruit and vegetable intake.There is no minimum or maximum available for this measure.
  The frequency reported categorically on the questionnaire was converted to the number of times fruits/vegetables were consumed per day as shown below. In general, the midpoint of the frequency range was used.
  Frequency ResponseTimes Per Day Never 0.0 Less than once a month 0.018 1-3 times per month 0.066 1-2 times per week 0.214 3-4 times per week 0.499 5-6 times per week 0.784
  1. time per day 1.0
  2. or more times per day 2.0
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: Times fruit/vegetable consumed per day
Arm/Group | Intervention
Number analyzed (Participants) | 12
Times fruit/vegetable consumed per day
  T1 (baseline) | 4.87 (3.42)
  T2 (post-intervention) | 5.72 (3.43)
  T2 vs. T1 | 0.85 (1.75)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.32 to 2.03]

5. Secondary Outcome: Frequency of Added Sugar Intake
Description: NCI brief Added Sugar intake survey was used to measure dietary intake. Participants reported the frequency of each specific food eaten over the past 12 months. Values are:1 = never, 2 = less than once per month,3 = 1-3 times per week, 4 = 3-4 times per week,5 = 5-6 times per week, 6 = 1 time per day, 7 = 2 or more times per day. Higher scores indicate more frequent fat intake.There is no minimum or maximum available for this measure.
  The frequency reported categorically on the questionnaire was converted to the number of times consumed per day as shown below. In general, the midpoint of the frequency range was used.
  Frequency ResponseTimes Per Day Never 0.0 Less than once a month 0.018 1-3 times per month 0.066 1-2 times per week 0.214 3-4 times per week 0.499 5-6 times per week 0.784
  1. time per day 1.0
  2. or more times per day 2.0
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: Times added sugar consumed per day
Arm/Group | Intervention
Number analyzed (Participants) | 12
Times added sugar consumed per day
  T1 (baseline) | 21.07 (14.88)
  T2 (post-intervention) | 12.53 (8.32)
  T2 vs. T1 | -8.54 (17.88)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = -0.48, t-test, 2 sided; Mean Difference (Final Values) = -8.54, 95% CI 2-sided [-19.9 to 2.82]

6. Secondary Outcome: Daily Physical Activity (Metabolic Equivalent Task MET)
Description: The International Physical Activity Questionnaire Short Form (7 items) was be used to measure physical activity. Participants are asked to report frequency (days/week) and duration (hours/ day or minutes/day) of vigorous and moderate physical activities performed in the past 7 days.
  Participants were asked about 3 specific types of activity: walking, moderate-intensity activity, and vigorous-intensity activity. Participants also reported frequency (days per week) and duration (time per day) for each specific type of activity. To create metabolic equivalent of task (MET, energy expenditure) measures, we multiplied frequency by duration (in hours). We then used the summation times 3.3 MET (walking), 4.0 (moderate physical activity), and 8.0 (vigorous physical activity) to generate physical activity scores in MET units. Higher scores indicated more energy expenditure.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: MET - Minutes per week
Arm/Group | Intervention
Number analyzed (Participants) | 12
MET - Minutes per week
  T1 (baseline) | 107.0 (249.6)
  T2 (post-interveion) | 171.5 (390.0)
  T2 vs. T1 | 64.46 (504.1)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = 64.46, 95% CI 2-sided [-256 to 384.7]

7. Secondary Outcome: Change in Autonomous Motivation for Stress Management
Description: Autonomous motivation. To measure autonomous motivation, we used the Treatment Self-Regulation Questionnaire (6 items for stress management). Participants rated how true each statement was for them related to stress management using a 7-point scale: 1 (not at all true) to 7 (very true). We summed responses to the 6 items to create a score for stress management. Scores can range from 6 - 42. Higher scores indicated higher autonomous motivation.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 36.50 (4.87)
  T2 (post-intervention) | 40.00 (2.83)
  T2 vs. T1 | 3.50 (3.97)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.88, t-test, 2 sided; Mean Difference (Final Values) = 3.50, 95% CI 2-sided [0.98 to 6.02]

8. Secondary Outcome: Change in Autonomous Motivation for Healthy Eating
Description: Autonomous motivation. To measure autonomous motivation, we used the Treatment Self-Regulation Questionnaire (6 items for healthy eating). Participants rated how true each statement was for them related to healthier eating using a 7-point scale: 1 (not at all true) to 7 (very true). We summed responses to the 6 items to create a score for healthy eating. Scores can range from 6 - 42 Higher scores indicated higher autonomous motivation.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 37.58 (4.01)
  T2 (post-intervention) | 40.25 (3.22)
  T2 vs. T1 | 2.67 (3.58)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [-0.10 to 4.94]

9. Secondary Outcome: Change in Autonomous Motivation for Physical Activity
Description: Autonomous motivation. To measure autonomous motivation, we used the Treatment Self-Regulation Questionnaire (6 items for physical activity). Participants rated how true each statement was for them related to physical activity using a 7-point scale: 1 (not at all true) to 7 (very true). We summed responses to the 6 items to create a score for physical activity. Scores can range from 6 -42. Higher scores indicated higher autonomous motivation.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 36.00 (5.72)
  T2 (post-intervention) | 40.50 (2.71)
  T2 vs. T1 | 4.50 (5.79)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.78, t-test, 2 sided; Mean Difference (Final Values) = 4.50, 95% CI 2-sided [0.82 to 8.18]

10. Secondary Outcome: Change in General Self-efficacy
Description: Self-efficacy. We used surveys to measure self-efficacy. We also used the general self-efficacy scale (10 items) to measure self-efficacy. Participants rated the truthfulness of each statement using a 4-point scale: 1 (not at all true) to 4 (exactly true). We summed responses to the 10 items to create a score for general self-efficacy. Scores can range from 10 - 40. Higher scores meant higher self-efficacy.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 31.42 (5.18)
  T2 (post-intervention) | 34.83 (4.24)
  T2 vs. T1 | 3.42 (5.88)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.58, t-test, 2 sided; Mean Difference (Final Values) = 3.42, 95% CI 2-sided [-0.32 to 7.16]

11. Secondary Outcome: Change in Healthy Eating Self-efficacy
Description: Self-efficacy. We used surveys to measure self-efficacy for healthy eating (8 items). Participants rated levels of confidence using a 4-point scale: 1 (not at all confident) to 4 (very confident). We summed responses to the 8 items to create a score for self-efficacy for healthy eating. THigher scores meant higher self-efficacy. Participants rated the truthfulness of each statement using a 4-point scale: 1 (not at all true) to 4 (exactly true). We summed responses to the 10 items to create a score for general self-efficacy.
  Scores can range from 8 - 32. Higher scores meant higher self-efficacy.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 19.83 (4.90)
  T2 (post-intervention) | 22.25 (4.88)
  T2 vs. T1 | 2.42 (3.96)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 2.42, 95% CI 2-sided [-0.10 to 4.94]

12. Secondary Outcome: Change in Physical Activity Self-efficacy
Description: Self-efficacy. We used surveys to measure physical activity (10 items). Participants rated levels of confidence using a 4-point scale: 1 (not at all confident) to 4 (very confident). We summed responses to the 10 items to create a score for self-efficacy for physical activity. Higher scores meant higher self-efficacy. Participants rated the truthfulness of each statement using a 4-point scale: 1 (not at all true) to 4 (exactly true). We summed responses to the 10 items to create a score for general self-efficacy. Scores can range from 10 - 40. Higher scores meant higher self-efficacy.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 25.33 (7.18)
  T2 (post-intervention) | 29.17 (7.41)
  T2 vs. T1 | 3.83 (8.39)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.46, t-test, 2 sided; Mean Difference (Final Values) = 3.83, 95% CI 2-sided [-1.50 to 9.16]

13. Secondary Outcome: Change in Emotion Regulation
Description: Emotional control. To measure emotional control, we used the Emotion Regulation Questionnaire to assess the emotional regulatory process using reappraisal (6 items) and suppression (4 items). Participants rated the degree of agreement using a 7-point scale: 1 (strongly disagree) to 7 (strongly agree). The suppression items were reverse coded prior to score computation. We summed responses to the 10 items to create a score for emotional control. Scores could range between 10 - 70. Higher scores meant better emotional control.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
units on a scale
  T1 (baseline) | 38.50 (8.34)
  T2 (post-intervention) | 42.58 (10.61)
  T2 vs. T1 | 4.08 (5.74)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 4.08, 95% CI 2-sided [0.43 to 7.73]

14. Secondary Outcome: Change in Perceived Stress
Description: We used the Perceived Stress Scale (10 items) to measure stress. Participants rated the frequency of stressful life situations in the past month using a 4-point scale: 1 (never) to 4 (often). We summed responses to the 10 items to create a score for stress. Scores can range from 10-40. Higher scores meant perceived higher levels of stress.
Time Frame: baseline (T1) and 3 weeks follow up (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 12
score on a scale
  T1 (baseline) | 18.33 (6.10)
  T2 (post-inbtervention) | 14.67 (6.64)
  T2 vs. T1 | -3.67 (7.01)
Statistical Analysis 1: Comparison: Intervention; Test type: Non-Inferiority — Paired T test (pre- post-); p = -0.52, t-test, 2 sided; Mean Difference (Final Values) = -3.67, 95% CI 2-sided [-8.12 to 0.79]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT04649047/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04649047/ICF_001.pdf